CLINICAL TRIAL: NCT01585558
Title: Long-Term Safety of 30 mg and 60 mg Oral Daily Dose of Ospemifene in the Treatment of Vulvar and Vaginal Atrophy (VVA) in Postmenopausal Women With Intact Uterus: A 40 Week Randomized, Double Blind, Placebo Controlled, Follow-Up to Protocol 15-50310.
Brief Title: Long-Term Safety of 30 mg and 60 mg Oral Daily Dose of Ospemifene in the Treatment of Vulvar and Vaginal Atrophy (VVA) in Postmenopausal Women With Intact Uterus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Collaborators: QuatRx Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-50310X
Record Dates: First submitted 2012-04-18; First posted 2012-04-26 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-04

CONDITIONS: Atrophy; Vaginal Diseases
Keywords: Menopausal symptoms; Urogenital atrophy; Vulvar and vaginal atrophy in menopausal women; Vaginal atrophy
MeSH Terms: conditions — Atrophy; Vaginal Diseases | interventions — Ospemifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Treatment Group 1 (Experimental)
  Interventions: Drug: Ospemifene (Dose 1)
- Treatment Group 2 (Experimental)
  Interventions: Drug: Ospemifene (Dose 2)
- Treatment Group 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ospemifene (Dose 1)
  Arms: Treatment Group 1
Drug: Ospemifene (Dose 2)
  Arms: Treatment Group 2
Drug: Placebo
  Arms: Treatment Group 3

SUMMARY:
The primary objective of the study was to assess the long-term safety of 30- and 60-mg daily doses of ospemifene in the treatment of Vulvar and Vaginal Atrophy (VVA) in postmenopausal women with an intact uterus.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 40 to 80 years with a diagnosis of vulvar and vaginal atrophy (VVA) as assessed by vaginal pH, maturation index of vaginal smear, and self-reported symptoms at Baseline for Protocol 15-50310
* Had an intact uterus
* Met the inclusion and exclusion criteria for Protocol 15-50310
* Had completed Protocol 15-50310

Exclusion Criteria:

* Had clinically significant abnormal findings at the Week 12 End of Study visit for Protocol 15-50310
* Had any physical or mental condition which, in the opinion of the investigator, may have interfered with the subject's ability to comply with the study procedures

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2006-05-16 (Actual); Primary Completion 2008-08-19 (Actual); Study Completion 2008-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi

REFERENCES:
- [Derived] Lara LA, Cartagena-Ramos D, Figueiredo JB, Rosa-E-Silva ACJ, Ferriani RA, Martins WP, Fuentealba-Torres M. Hormone therapy for sexual function in perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2023 Aug 24;8(8):CD009672. doi: 10.1002/14651858.CD009672.pub3. PMID 37619252

RESULTS

PARTICIPANT FLOW:
Groups:
- Ospemifene 30 mg (Dose 1): Subjects took a daily oral dose of one 30 mg ospemifene film-coated tablet each morning with food for 40 weeks
- Ospemifene 60 mg (Dose 2): Subjects took a daily oral dose of one 60 mg ospemifene film-coated tablet each morning with food for 40 weeks
- Placebo: Subjects took a daily oral dose of one placebo tablet (identical in appearance to ospemifene tablets) each morning with food for 40 weeks
Period: Overall Study
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Started | 62 | 69 | 49
Completed | 49 | 57 | 34
Not Completed | 13 | 12 | 15
Not completed — Withdrawal by Subject | 4 | 5 | 8
Not completed — Lost to Follow-up | 2 | 0 | 3
Not completed — Adverse Event | 3 | 4 | 1
Not completed — Protocol Violation | 4 | 3 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo | Total
Number analyzed (Participants) | 62 | 69 | 49 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (6.13) | 57.7 (5.88) | 58.2 (4.02) | 58.1 (5.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 69 | 49 | 180
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 6
  Not Hispanic or Latino | 61 | 66 | 47 | 174
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 58 | 61 | 43 | 162
  Black or African American | 4 | 4 | 2 | 10
  Asian | 0 | 2 | 1 | 3
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Other | 0 | 1 | 2 | 3
  Missing value | 0 | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: cm] | 162.83 (6.930) | 162.53 (6.488) | 163.27 (6.082) | 162.84 (6.509)
Weight [Mean (Standard Deviation); unit: kg] | 68.92 (11.316) | 65.52 (11.626) | 66.71 (10.482) | 67.02 (11.252)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.014 (4.1507) | 24.792 (4.1292) | 25.045 (3.8496) | 25.282 (4.0762)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Time Frame: Week 20 (Phone Contact) to Week 56 (Visit 7)
Measure: Number; unit: Participants
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 62 | 69 | 49
Participants
  Treatment-Emergent AE | 38 | 44 | 22
  Related AE (Possibly/Probably/Definitely Related) | 11 | 18 | 5
  AE Causing Study Drug Discontinuation | 3 | 4 | 1
  Serious AE | 2 | 5 | 1
  Severe AE | 6 | 7 | 2

2. Primary Outcome: Assessment of Cervical Pap Smear Samples
Description: Cervical Pap smear samples were used to evaluate: atypical squamous cells of undetermined significance (ASC-US), squamous intraepithelial lesions (SILs), intraepithelial lesions or malignancy, and reactive endocervical cells and/or metaplastic cells.
Time Frame: Week 52 (Visit 6)
Population: The ITT population was used for the analysis. For this particular outcome measure, 49 out of 62 subjects in the ospemifene 30 mg group, 58 out of 69 subjects in the ospemifene 60 mg group, and 34 out of 49 subjects in the placebo group were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 34
Participants
  ASC-US | 1 | 2 | 0
  Inadequate squamous epithelial component | 1 | 0 | 1
  Low grade SIL (slight dysplasia and/or HPV effect) | 0 | 1 | 0
  Negative for intraepithelial lesion or malignancy | 45 | 54 | 33
  Reactive endocervical and/or metaplastic cells | 1 | 1 | 0
  Unsatisfactory: Due to reasons noted | 1 | 0 | 0

3. Primary Outcome: Assessment of Endometrial Biopsy
Description: Assessments were based on Blaustein's classification.
Time Frame: Week 52 (Visit 6)
Population: The ITT population was used for the analysis. For this particular outcome measure, at Week 52, 46 out of 62 subjects in the ospemifene 30 mg group, 55 out of 69 subjects in the ospemifene 60 mg group, and 32 out of 49 subjects in the placebo group were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 46 | 55 | 32
Participants
  Atrophic/inactive/insufficient | 44 | 53 | 32
  Weakly proliferative | 1 | 1 | 0
  Atypical epithelial proliferation | 1 | 0 | 0
  Proliferative pattern, disordered type | 0 | 1 | 0
  Other (Polyp, atrophic type) | 0 | 0 | 0
  Hyperplasia or carcinoma | 0 | 0 | 0

4. Primary Outcome: Mean Percent Change From Baseline in Serum Lipids
Time Frame: Baseline to Week 26 (Visit 5)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 62 | 69 | 49
percent change
  Total Cholesterol | -0.14 (14.807) | 2.35 (13.663) | 6.24 (12.904)
  Low-density-lipoprotein cholesterol (LDL-C) | -0.02 (19.462) | 2.42 (19.107) | 10.38 (19.776)
  High-density-lipoprotein cholesterol (HDL-C) | 6.48 (13.881) | 5.76 (12.686) | 2.39 (14.026)
  Triglycerides | -0.66 (28.864) | 5.12 (31.076) | 20.36 (41.755)

5. Primary Outcome: Mean Percent Change From Baseline in Serum Lipids
Time Frame: Baseline to Week 52 (Visit 6)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 62 | 69 | 49
percent change
  Total Cholesterol | -0.55 (13.910) | -2.45 (12.323) | -1.05 (9.289)
  LDL-C | -0.87 (19.748) | -6.20 (18.623) | -0.42 (15.418)
  HDL-C | 6.07 (16.836) | 1.29 (12.787) | -4.41 (14.347)
  Triglycerides | -3.10 (32.749) | 15.19 (35.789) | 21.57 (40.802)

6. Primary Outcome: Mean Change in Blood Chemistry Parameters
Time Frame: Baseline to Week 26 (Visit 5)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 62 | 69 | 49
U/L
  Alanine Aminotransferase (ALT) | -1.2 (9.39) | -1.3 (8.73) | -1.3 (8.22)
  Aspartate Aminotransferase (AST) | 0.8 (4.67) | 1.2 (5.43) | 0.5 (4.59)
  Creatine Kinase (CK) | 1.1 (50.97) | -4.4 (48.78) | 18.7 (69.50)

7. Primary Outcome: Mean Change in Blood Chemistry Parameters
Time Frame: Baseline to Week 52 (Visit 6)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 62 | 69 | 49
U/L
  ALT | -2.1 (10.27) | -3.2 (7.91) | -2.2 (7.21)
  AST | 1.5 (4.99) | 0.5 (5.03) | 0.3 (4.95)
  CK | 7.3 (62.70) | 1.2 (56.78) | -6.0 (31.82)

8. Primary Outcome: Assessment of Endometrial Safety With a Transvaginal Ultrasound (TVU)
Description: Mean change in endometrial thickness from baseline
Time Frame: Baseline to Week 26 (Visit 5)
Population: The ITT population was used for the analysis. For this particular outcome measure, at Week 26, 50 out of 62 subjects in the ospemifene 30 mg group, 60 out of 69 subjects in the ospemifene 60 mg group, and 37 out of 49 subjects in the placebo group were analyzed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 50 | 60 | 37
mm | 0.580 (1.9041) | 0.818 (1.6689) | -0.119 (1.1629)

9. Primary Outcome: Assessment of Endometrial Safety With a TVU
Description: Mean change in endometrial thickness from baseline
Time Frame: Baseline to Week 52 (Visit 6)
Population: The ITT population was used for the analysis. For this particular outcome measure, at Week 52, 46 out of 62 subjects in the ospemifene 30 mg group, 52 out of 69 subjects in the ospemifene 60 mg group, and 30 out of 49 subjects in the placebo group were analyzed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 46 | 52 | 30
mm | 0.681 (2.5666) | 1.139 (1.5568) | -0.041 (1.1455)

10. Primary Outcome: Change From Baseline in Visual Evaluation of the Vagina
Description: Petechiae, pallor, friability, dryness in the mucosa, and redness in the mucosa were assessed on a 4-point scale (0=None, 1=Mild, 2=Moderate, 3=Severe).
Time Frame: Baseline to Week 26 (Visit 5)
Population: The ITT population was used for the analysis. For this particular outcome measure, at Week 26, 52 out of 62 subjects in the ospemifene 30 mg group, 65 out of 69 subjects in the ospemifene 60 mg group, and 42 out of 49 subjects in the placebo group were analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 65 | 42
Units on a scale
  Petechiae | -0.7 (0.94) | -0.6 (0.82) | -0.3 (0.79)
  Pallor | -1.3 (0.89) | -1.2 (1.02) | -0.5 (0.94)
  Friability | -0.9 (1.02) | -0.8 (0.95) | -0.6 (0.99)
  Vaginal Dryness in Mucosa | -1.6 (1.07) | -1.4 (0.91) | -0.8 (1.11)
  Vaginal Redness in Mucosa | -0.8 (0.96) | -0.7 (0.95) | -0.4 (0.89)

11. Primary Outcome: Change From Baseline in Visual Evaluation of the Vagina
Description: as for outcome 10
Time Frame: Baseline to Week 52 (Visit 6)
Population: The ITT population was used for the analysis. For this particular outcome measure, at Week 52, 49 out of 62 subjects in the ospemifene 30 mg group, 58 out of 69 subjects in the ospemifene 60 mg group, and 35 out of 49 subjects in the placebo group were analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
Units on a scale
  Petechiae | -0.8 (0.85) | -0.7 (0.91) | -0.4 (0.73)
  Pallor | -1.3 (0.74) | -1.2 (1.15) | -0.6 (1.03)
  Friability | -0.9 (0.91) | -0.7 (0.95) | -0.5 (0.92)
  Vaginal Dryness in Mucosa | -1.7 (0.96) | -1.4 (1.06) | -1.1 (1.02)
  Vaginal Redness in Mucosa | -0.8 (0.96) | -0.6 (1.03) | -0.5 (1.07)

12. Primary Outcome: Change From Baseline in Estradiol (E2) Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: The ITT population was used for the analysis. For this particular outcome measure, at Week 26, 52 out of 62 subjects in the ospemifene 30 mg group, 63 out of 69 subjects in the ospemifene 60 mg group, and 42 out of 49 subjects in the placebo group were analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
pg/mL | 0.75 (3.27) | 0.94 (5.97) | 0.15 (0.79)

13. Primary Outcome: Change From Baseline in Luteinizing Hormone (LH) Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
IU/L | -2.02 (5.26) | -2.86 (6.97) | -0.83 (4.82)

14. Primary Outcome: Change From Baseline in Follicle Stimulating Hormone (FSH) Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
IU/L | -7.44 (11.78) | -9.87 (14.00) | -4.10 (11.37)

15. Primary Outcome: Change From Baseline in Sex Hormone Binding Globulin (SHBG) Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
nmol/L | 11.71 (19.64) | 22.64 (28.07) | -2.74 (12.84)

16. Primary Outcome: Change From Baseline in Testosterone (Total) Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
ng/dL | 1.61 (5.29) | 2.59 (5.75) | -0.76 (7.18)

17. Primary Outcome: Change From Baseline in Testosterone (Free) Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
ng/dL | -0.01 (0.13) | -0.00 (0.22) | -0.03 (0.15)

18. Primary Outcome: Change From Baseline in E2 Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
pg/mL | 0.06 (1.27) | -0.02 (1.05) | 0.14 (0.69)

19. Primary Outcome: Change From Baseline in LH Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
IU/L | -2.65 (6.73) | -4.95 (7.59) | -0.09 (5.45)

20. Primary Outcome: Change From Baseline in FSH Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
IU/L | -12.39 (16.88) | -15.60 (13.32) | -6.29 (17.39)

21. Primary Outcome: Change From Baseline in SHBG Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
nmol/L | 11.94 (20.81) | 28.09 (25.62) | -5.94 (13.33)

22. Primary Outcome: Assessment of Mammography
Description: Mammography was done for the detection of characteristic masses and microcalcifications in the breast.
Time Frame: Week 52 (Visit 6)
Measure: Number; unit: Participants
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 62 | 69 | 49
Participants
  Breast cyst | 0 | 0 | 1
  Breast mass | 2 | 1 | 0
  Breast microcalcification | 0 | 1 | 0
  Mammogram abnormal | 0 | 1 | 0

23. Primary Outcome: Change From Baseline in Testosterone (Total) Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
ng/dL | 1.92 (5.13) | 3.48 (7.86) | -0.95 (4.60)

24. Primary Outcome: Change From Baseline in Testosterone (Free) Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
ng/dL | 0.02 (0.10) | -0.01 (0.15) | 0.01 (0.12)

25. Primary Outcome: Change From Baseline in Antithrombin Antigen, P Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
percent change | 0.7 (10.15) | -2.4 (11.23) | 1.2 (10.49)

26. Primary Outcome: Change From Baseline in Fibrinogen Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
mg/dL | -29.1 (83.18) | -25.9 (63.17) | 12.1 (70.52)

27. Primary Outcome: Change From Baseline in Protein C Ag, P Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
percent change | 8.2 (20.20) | -2.0 (20.68) | 14.2 (21.96)

28. Primary Outcome: Change From Baseline in Protein S Ag (Free), P Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
percent change | 4.7 (13.33) | 6.8 (12.82) | 4.8 (9.79)

29. Primary Outcome: Change From Baseline in Thromboplastin Time
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 63 | 42
s | 0.5 (7.48) | -0.6 (3.37) | 0.3 (2.87)

30. Primary Outcome: Change From Baseline in Antithrombin Antigen, P Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
percent change | 5.1 (9.56) | 1.0 (9.28) | 7.1 (11.64)

31. Primary Outcome: Change From Baseline in Fibrinogen Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
mg/dL | -24.0 (61.79) | -36.0 (67.82) | 7.4 (96.67)

32. Primary Outcome: Change From Baseline in Protein C Ag, P Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
percent change | 4.9 (17.11) | -2.9 (19.20) | 10.6 (20.11)

33. Primary Outcome: Change From Baseline in Protein S Ag (Free), P Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
percent change | 7.1 (16.77) | 11.1 (13.78) | 9.3 (15.92)

34. Primary Outcome: Change From Baseline in Thromboplastin Time
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
s | 0.4 (4.13) | 0.5 (3.43) | 1.2 (5.05)

35. Primary Outcome: Assessment of Breast Palpation
Description: Breast palpation was done by the investigator to assess abnormalities in the breast.
Time Frame: Week 26 (Visit 5)
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 65 | 42
Participants
  Not done | 0 | 1 | 0
  Normal | 52 | 64 | 41
  Abnormal | 0 | 0 | 1

36. Primary Outcome: Assessment of Breast Palpation
Description: Breast palpation was done by the investigator to assess abnormalities in the breast.
Time Frame: Week 52 (Visit 6)
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
Participants
  Normal | 49 | 57 | 35
  Abnormal | 0 | 1 | 0

37. Primary Outcome: Assessment of Hematology Tests
Description: Change from baseline
Time Frame: Baseline to Week 26 (Visit 5)
Population: The ITT population was used for the analysis. For this particular outcome measure, at Week 26, 51 out of 62 subjects in the ospemifene 30 mg group, 61 out of 69 subjects in the ospemifene 60 mg group, and 42 out of 49 subjects in the placebo group were analyzed.
Measure: Mean (Standard Deviation); unit: (x10(9)/L)
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 51 | 61 | 42
(x10(9)/L)
  Leukocytes (WBC) | -0.008 (1.2147) | -0.211 (1.3608) | 0.207 (1.0489)
  Basophils | 0.006 (0.0240) | 0.001 (0.0215) | -0.005 (0.0186)
  Lymphocytes | -0.035 (0.3169) | -0.064 (0.4004) | 0.116 (0.4972)
  Monocytes | 0.025 (0.1297) | -0.042 (0.1127) | 0.009 (0.1362)
  Neutrophils | -0.010 (0.9812) | -0.094 (1.2380) | 0.083 (0.7953)
  Eosinophils | -0.010 (0.0955) | -0.009 (0.1072) | 0.002 (0.1168)
  Platelet Count | -5.2 (31.23) | -5.6 (30.53) | -4.5 (31.56)

38. Primary Outcome: Change From Baseline in Erythrocyte (RBC) Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: (x10(12)/L)
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 51 | 61 | 42
(x10(12)/L) | -0.081 (0.2232) | -0.089 (0.2500) | 0.026 (0.2240)

39. Primary Outcome: Change From Baseline in Hemogobin Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 51 | 61 | 42
g/dL | -0.150 (0.6664) | -0.165 (0.6668) | 0.140 (0.6247)

40. Primary Outcome: Change From Baseline in Hematocrit Levels
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 51 | 61 | 42
percent change | -0.435 (2.0189) | -0.529 (2.1667) | 0.398 (1.9951)

41. Primary Outcome: Assessment of Hematology Test Values
Description: Change from baseline
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: (x10(9)/L)
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
(x10(9)/L)
  Leukocytes (WBC) | 0.061 (1.7480) | -0.217 (0.9597) | 0.371 (1.3680)
  Basophils | 0.003 (0.0181) | 0.002 (0.0281) | -0.003 (0.0214)
  Lymphocytes | -0.120 (0.4796) | 0.001 (0.3339) | -0.028 (0.3352)
  Monocytes | -0.024 (0.1065) | -0.028 (0.1017) | 0.021 (0.1216)
  Neutrophils | 0.194 (1.7491) | -0.258 (0.9189) | 0.377 (1.3568)
  Eosinophils | -0.003 (0.1029) | -0.005 (0.0823) | 0.021 (0.1889)
  Platelet Count | -11.2 (34.86) | -16.4 (27.80) | -11.3 (37.75)

42. Primary Outcome: Change From Baseline in Erythrocyte (RBC) Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: (x10(12)/L)
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
(x10(12)/L) | -0.087 (0.2115) | -0.155 (0.2113) | 0.028 (0.2350)

43. Primary Outcome: Change From Baseline in Hemoglobin Levels
Time Frame: Baseine to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
g/dL | -0.141 (0.6261) | -0.431 (0.6367) | 0.094 (0.6121)

44. Primary Outcome: Change From Baseline in Hematocrit Levels
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
percent change | -0.445 (1.9207) | -1.152 (1.9113) | 0.174 (2.0823)

45. Primary Outcome: Change From Baseline in pH of Urine
Time Frame: Baseline to Week 26 (Visit 5)
Population: The ITT population was used for the analysis. For this particular outcome measure, at Week 26, 52 out of 64 subjects in the ospemifene 30 mg group, 64 out of 69 subjects in the ospemifene 60 mg group, and 41 out of 49 subjects in the placebo group were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 64 | 41
pH | 0.2 (1.28) | 0.0 (0.97) | 0.1 (1.15)

46. Primary Outcome: Change From Baseline in Specific Gravtiy of Urine
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 64 | 41
units | -0.002 (0.0074) | -0.003 (0.0062) | -0.000 (0.0065)

47. Primary Outcome: Change From Baseline in pH of Urine
Time Frame: Baseline to Week 52 (Visit 6)
Population: The ITT population was used for the analysis. For this particular outcome measure, at Week 52, 49 out of 62 subjects in the ospemifene 30 mg group, 57 out of 69 subjects in the ospemifene 60 mg group, and 35 out of 49 subjects in the placebo group were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 57 | 35
pH | 0.1 (1.17) | 0.0 (1.15) | 0.2 (1.20)

48. Primary Outcome: Change From Baseline in Specific Gravity of Urine
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 57 | 35
units | -0.001 (0.0061) | -0.002 (0.0074) | -0.001 (0.0067)

49. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP)
Time Frame: Baseline to Week 26 (Visit 5)
Population: The ITT population was used for the analysis. For this particular outcome measure, at Week 26, 52 out of 62 subjects in the ospemifene 30 mg group, 66 out of 69 subjects in the ospemifene 60 mg group, and 42 out of 49 subjects in the placebo group were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 66 | 42
mmHg | -2.1 (15.33) | 2.4 (12.16) | 0.5 (11.16)

50. Primary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP)
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 66 | 42
mmHg | -2.0 (9.49) | 0.5 (8.29) | 0.3 (8.07)

51. Primary Outcome: Change From Baseline in Pulse Rate
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 66 | 42
bpm | 2.0 (11.71) | 0.8 (10.61) | 2.2 (8.60)

52. Primary Outcome: Change From Baseline in Weight
Time Frame: Baseline to Week 26 (Visit 5)
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 66 | 42
kg | -0.88 (3.902) | 0.66 (2.997) | 0.78 (2.732)

53. Primary Outcome: Change From Baseline in BMI
Time Frame: Baseline to Week 26
Population: as for outcome 49
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 52 | 66 | 42
kg/m^2 | -0.331 (1.4659) | 0.253 (1.1244) | 0.293 (1.0131)

54. Primary Outcome: Change From Baseline in SBP
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
mmHg | -4.5 (15.28) | 0.9 (15.30) | 4.2 (15.21)

55. Primary Outcome: Change From Baseline in DBP
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
mmHg | -2.5 (10.32) | 0.7 (9.97) | 0.8 (7.85)

56. Primary Outcome: Change From Baseline in Pulse Rate
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
bpm | 2.6 (9.78) | -0.5 (12.05) | 2.9 (6.61)

57. Primary Outcome: Change From Baseline in Weight
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
kg | -0.99 (4.975) | 0.98 (3.055) | 1.99 (3.084)

58. Primary Outcome: Change From Baseline in BMI
Time Frame: Baseline to Week 52 (Visit 6)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Number analyzed (Participants) | 49 | 58 | 35
kg/m^2 | -0.379 (1.8594) | 0.376 (1.1942) | 0.748 (1.1672)

ADVERSE EVENTS:
Time Frame: 40 weeks
Arm/Group | Ospemifene 30 mg (Dose 1) | Ospemifene 60 mg (Dose 2) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/62 | 5/69 | 1/49
Other Adverse Events (participants affected / at risk) | 9/62 | 21/69 | 11/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ospemifene 30 mg (Dose 1) (N=62) | Ospemifene 60 mg (Dose 2) (N=69) | Placebo (N=49)
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0
Encephalitis Herpes (Infections and infestations) | 0 | 1 | 0
Meningitis Candida (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast Cancer In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Breast Prosthesis Implantation (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ospemifene 30 mg (Dose 1) (N=62) | Ospemifene 60 mg (Dose 2) (N=69) | Placebo (N=49)
Nasopharyngitis (Infections and infestations) | 0 | 1 | 3
Sinusitis (Infections and infestations) | 4 | 2 | 2
Urinary Tract Infection (Infections and infestations) | 5 | 6 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 4 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Hot Flush (Vascular disorders) | 2 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.